CLINICAL TRIAL: NCT04727593
Title: The Modulatory Role of Internet-supported Mindfulness-based Cognitive Therapy on Extracellular Vesicles and Psychological Distress in People Who Have Had Cancer: A Study Protocol for a Two-armed Randomized Controlled Trial
Brief Title: The Modulatory Role of Internet MBCT on Extracellular Vesicles and Distress in Cancer Patients - Study Protocol
Acronym: MINDGAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Collaborators: European Commission (Other); University of Coimbra (Other); VTT Technical Research Centre, Finland (Other); University of Oulu (Other); Linnaeus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPO/PI134b
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Cancer; Internet; Extracellular vesicles; Distress; Mindfulness; Mindfulness Based Cognitive Therapy; Anxiety; Depression; Biomarkers; eHealth; Telehealth
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Masking Description: At baseline, everyone (participants, study coordinator, mindfulness instructor(s), research assistant, and statistician) will be blinded to conditions as it is expected to occur before randomization. Once participants are randomized, the study coordinator will inform them of the group assignments, and all of them will become unblinded to the conditions. Due to the specificities of this type of study and intervention, it is not possible to guarantee the blinding of personnel and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (MBCT) (Experimental): Group intervention on Mindfulness-Based Cognitive Therapy classic program plus 4 monthly consolidation sessions of 90 minutes each.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
- Treatment as Usual (TAU) (Other): TAU will be the control condition.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy (MBCT) — Experimental group: MBCT is program developed by Zindel Segal, Mark Williams, and John Teasdale , based on Jon Kabat-Zinn's Mindfulness-based Stress Reduction (MBSR) program. Participants learn to acknowledge their unhelpful thoughts and feelings, allowing the mind to move from an automatic and spiraling thought pattern to a more conscious emotional processing. Mindfulness practices include breath awareness, sitting and walking meditations, and mindful yoga. In this study, the following MBCT structure will be followed: group setting of 12 participants (maximum); 8 online weekly meetings of 2 hours via a videoconference platform (e.g., Cisco Webex), each one mediated by a trained mindfulness instructor(s); daily home practice of the learned skills; 2 hours of retreat after the fifth week; 6 months of home practice; 4 monthly consolidation sessions of 90 minutes each.
  Arms: Mindfulness Based Cognitive Therapy (MBCT)
Other: Treatment as Usual — In this case, participants will follow the usual institutional intervention protocol for medical follow-up and identification, referral, and intervention for people with significant distress difficulties. Regarding pharmacological intervention, medication intake will be monitored during the study and changes will be registered. The engagement in non-pharmacological interventions such as psychological and psychosocial interventions will also be monitored.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Mindfulness-based interventions (MBIs), such as mindfulness-based stress reduction (MBSR), mindfulness-based cognitive therapy (MBCT), mindfulness-based cancer recovery (MBCR), have been showing promising results in different health-related and psychosocial outcomes in the context of cancer. More recently, the possibility of delivering MBIs using technological tools and resources, such as internet and applications, has been receiving much attention, also accompanied by promising findings. However, few randomized controlled studies have been conducted and published to date. Moreover, few studies have addressed the long-term stability and trajectory of gains across time. Also, even though prior evidence had suggested that face-to-face MBIs might modulate several biological markers (e.g., pro-inflammatory gene expression and inflammatory signaling; telomere length), as far as we know, no previous study addressed the impact of online MBIs on biological indices, especially on extracellular vesicles (EVs).

As primary objective, this study aims to investigate the effects of an internet-based MBCT intervention (vs. Treatment as Usual - TAU) on EVs (objective measure), as well as on psychological distress (subjective measure), considering a sample of distressed people with history of breast, prostate, and colorectal cancer.

As secondary objective, this study aims to investigate the effects of this same intervention on psychosocial outcomes, including quality of life, fear of cancer recurrence, emotion suppression, mindfulness, sleep quality, posttraumatic growth, health-related behaviours (physical activity; smoking habits), and perceived social support. The biological secondary outcomes studied will be: inflammatory response genes interleukins (ILs, IL-1, IL-6, IL-8, IL-10), interferon gamma (IFN-γ), tumour necrosis factor (TNF), and c-reactive protein (CRP); telomerase activity; antigens related to cancer (cancer antigen - CA 15-3; prostate-specific antigen - PSA; carcinoembryonic antigen - CEA); other health-related markers (adrenocorticotropic hormone - ACTH; erythrocytes number; hemoglobin glycosylated).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast, prostate, or colorectal cancer;
* Cancer stage I - III;
* Primary cancer treatments completed between 3 months and 5 years (participants with ongoing adjuvant hormonal therapies will be included);
* Age between 18 and 65 years;
* Experiencing significant distress on the Distress Thermometer (DT ≥ 4)
* Willingness to accept randomization to one of the two study conditions and to attend the study for its duration;
* Ability to speak, read, and write in Portuguese and literacy to complete autonomously the self-report measures;
* Sufficient digital literacy with access to a device (e.g., smartphone; tablet; computer) with camera, microphone, and internet.

Exclusion Criteria:

* Concurrent diagnosis of severe psychiatric condition(s) (e.g., psychosis; substance abuse; bipolar disorder; suicidal ideation);
* Concurrent diagnosis of autoimmune disorder;
* Current use of antipsychotics;
* Current use of anti-inflammatory medication (corticotherapy);
* Undergoing trastuzumab therapy;
* Participation in a structured mindfulness program (e.g., MBCT; MBSR; Mindfulness-Based Cancer Recovery - MBCR) program in the past five years;
* Currently attending psychological consultation;
* Being pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change on Extracellular Vesicles | T1 - before intervention; 8 weeks after T1; 24 weeks after T1
  Isolated by ultracentrifugation with sucrose cushion. The collected EVs will be quantified by Nanoparticle tracking analysis (Nanosight Ltd.), and data will be measured in particles per milliliter (mL).
Change on Distress | T1- before intervention; T2 - 4 weeks after baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with Depression Anxiety Stress Scales-21 - DASS-21, a self-report and public domain questionnaire that evaluates negative affective states. It is composed of 21 items, 7 focused on depression, 7 on anxiety, and 7 on stress. Each item is rated on a 4-point Likert-type scale, wherein in 0 represents "did not apply to me at all" and 3 represents "applied to me very much or most of the time". The score for each subscale ranges between 0 and 21. In the current study, a total score will be computed by summing all items, with higher scores being indicative of higher self-reported psychological distress.

SECONDARY OUTCOMES:
Change on Cancer antigen 15-3 (CA 15-3) | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  Using an immunoassay analyser (units/mL).
Change on Prostate-specific antigen (PSA) | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  Using an immunoassay analyser (ng/mL).
Change on Carcinoembryonic Antigen (CEA). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  Using an immunoassay analyser (ng/mL).
Change on Adrenocorticotropic Hormone (ACTH). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  Using an immunoassay analyser (pg/mL).
Transcript inflammatory response genes (Interleukins, ILs, IL-1, IL-6, IL-8, IL-10, IFNγ and TNF). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  Assessed by quantitative RT-PCR (TaqMan™ Gene Expression Assays).
Change on Analytic biomarkers (Erythrocyte number). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  This indicator assesses erythrocytes number (million/mm3) from blood samples (Sysmex XN).
Change on Analytic biomarkers (PCR number). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  This indicator assesses PCR (mg/L) from blood samples.
Change on Analytic biomarkers (telomerase activity). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  This indicator assesses telomerase activity (units) from blood samples.
Change on Analytic biomarkers (hemoglobin glycosylated). | T1- before intervention; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline
  This indicator assesses High Performance Liquid Chromatography - HPLC, (mmol/mol) from blood samples.
Change on Global distress | T0 - Screening; T2 - 4 weeks after baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with Clinical Outcome Routine Evaluation - Outcome Measure, (CORE-OM) , a self-report measure of global distress (GD), comprising 34 items and four domains: subjective well-being, commonly experienced problems or symptoms, social/life functioning, and risk to self and others. The measure is scored on a 5-point scale ranging from 0 ('not at all') to 4 ('all the time'). The measure is suitable for use across a wide range of settings, it has been validated in different adult population with mental health problems, and it is sensitive to change.
Change on quality of life | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured by World Health Organization Quality of Life - Bref - WHOQOL-Bref, a questionnaire suitable for epidemiological and clinical trials, which assesses quality of life as proposed by WHO. It is composed of 26 items distributed in one general facet and four domains (physical health, psychological, social relationships, and environment). Each item is rated on a 5-point Likert-type scale with higher scores being indicative of better self-reported quality of life (scoring procedures are available here: https://www.who.int/mental_health/media/en/76.pdf).
Change on fear of cancer recurrence | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured by a 7-item Fear of Cancer Recurrence - FCR-7 (PT version not yet available), a 7-item scale assessing fear of cancer recurrence in a 5-point Likert scale ranging from 1 (not at all) to 5 (all the time). It had demonstrated good psychometric properties. We will translate, adapt and validate this measure, following the usual procedures to adapt psychological measures.
Change on satisfaction perceived social support | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Satisfaction with Social Support Scale - SSSS, a 15-item scale assessing social support satisfaction discriminating four dimensions: satisfaction with friends/friendships, intimacy, satisfaction with family and social activities.
Change on emotional suppression | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Emotion Regulation Questionnaire - ERQ) , - Only the subscale of emotion suppression composed of 4-items will be used. The items are rated in 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Change on mindfulness abilities | T1 Baseline; T2 - 4 weeks after baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured by Mindfulness Five Facet Mindfulness Questionnaire - FFMQ, a 39 items questionnaire that assess mindfulness and self-awareness states in everyday life, which are organized in five different facets/subscales: observing, describing, acting with awareness, nonreactivity to inner experience, and nonjudging of inner experience. Each item is rated on a 5-point Likert-type scale ranging from 1 (never or very rarely true) and 5 (very often or always true).
Change Interview | T3 - 8 weeks after baseline
  This interview assesses the psychotherapeutic changes perceived by participants after psychological intervention. The interview questions explore the changes that a person has noticed since therapy began, what the person attributes these changes to, and helpful and unhelpful aspects of therapy, in a qualitative way.
Change on smoking dependency | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with Fageström Test for Nicotine Dependence - FTND. This instrument assesses nicotine dependency with 6 items (rated from 0 to 2 or 3). The total score range is 1-10, with higher values meaning higher nicotine dependency.
Change on physical activity | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with International Physical Activity Questionnaire - Short Form - IPAQ-SF. This instrument assesses physical activity in 7 items, with higher scores meaning higher level of physical activity.
Change on sleep quality | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with Basic Scale on Insomnia complaints and Quality of Sleep - BaSIQS - This is a self-report measure that focus on evaluating sleep quality, as well as problems to fall asleep and maintain sleep. It encompasses 7 items rated in a 5-point Likert-type and the total score ranges between 0 and 28, with highest values indicating poor sleep quality. Satisfactory psychometric properties were reported in the original study with Portuguese higher education students, but also on community and clinical samples
Change on posttraumatic growth | T1 - Baseline; T3 - 8 weeks after baseline; T4 - 24 weeks after baseline; T5 - 52 weeks after baseline
  Measured with Posttraumatic Growth Inventory - PTGI, which is a self-report questionnaire that evaluates positive psychological change in people experiencing traumatic events. It includes 21 items and each item is rated on a 6-point Likert-type scale ranging from 0 ("I did not experience this change as a result of my crisis") to 5 ("I experienced this change to a very great degree as a result of my crisis"). Total score ranges between 0 and 105, with higher values being indicative of a greater degree of posttraumatic growth.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Henrique, PhD, Study Director — Institute of Oncology of Porto, Portugal; Carmen Jerónimo, PhD, Study Director — Institute of Oncology of Porto, Portugal; Eunice Silva, PhD, Study Director — Institute of Oncology of Porto, Portugal
Locations (1):
- Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto, Portugal

REFERENCES:
- [Derived] Pereira DR, Silva ER, Carvalho-Maia C, Monteiro-Reis S, Lourenco C, Calisto R, Teixeira RJ, Carlson LE, Bart G, Vainio SJ, Sales MGF, Jeronimo C, Henrique R. The modulatory role of internet-supported mindfulness-based cognitive therapy on extracellular vesicles and psychological distress in people who have had cancer: a protocol for a two-armed randomized controlled study. Trials. 2022 Feb 5;23(1):118. doi: 10.1186/s13063-022-06045-x. PMID 35123569
- See also: MindGAP project website — http://mindgap-fet-open.eu/